CLINICAL TRIAL: NCT02062567
Title: Ultrasonographic Guided Treatment of Acute Achilles Tendon Rupture. Evaluation of Two Novel Ultrasonographic Measurements
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: DJO Incorporated (Industry); The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Kristoffer Barfod, MD, PhD, Hvidovre University Hospital
Other Study IDs: ATR_US_Denmark_2014
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Achilles Tendon; Rupture; Ultrasound
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Achilles tendon rupture

SUMMARY:
With this project the investigators wish to:

1. Test the reproducibility of Amlang's ultrasound classification by examining the intra- and inter-rater reliability.
2. Investigate whether Amlang's ultrasound classification is able to predict which patients are likely to develop complications when treated non-operatively.
3. Investigate whether Barfod's length measurement is able to predict which patients are likely to develop complications when treated non-operatively.

DETAILED DESCRIPTION:
Study objectives

To validate Amlang's ultrasound classification and investigate whether the treatment of acute Achilles tendon ruptures (ATR) can be guided by:

1. Amlang's ultrasound classification of ATR
2. Barfod's ultrasound measurement to determine the elongation of the Achilles tendon following a rupture Backgrund A larger group of patients end up with a poor outcome after treatment for ATR. ATR is a frequent and potentially debilitating injury that typically affects young active adults (11 to 37 per 100,000)1 2 3. Consequently, there are great socioeconomic benefits in optimizing treatment and shortening time of recovery.

There is currently no consensus regarding the best treatment of ATR. Traditionally the operative treatment has been considered superior, however recent studies show that non-operative treatment is a safe treatment which leads to good results 4 5 6. For this reason a transition towards greater use of non-operative treatment is seen in many orthopedic departments 7.

Patients who end up with a poor result after treatment for ATR typically suffer from rerupture of the tendon or an elongation of the tendon. There is a 5-10 percent risk of rerupture 4 5 6. It is unknown how many patients heal with an elongation of the Achilles tendon. Correct length of the Achilles tendon is essential for the subsequent function of the tendon.

In order to shorten time of recovery and optimize the treatment-outcome, it is desirable to identify patients at risk of re-rupture or elongation as early as possible as early surgery might help these patients.

Amlang et al. have developed an ultrasonographic classification system to be used in the acute phase of rupture 8. The aim is to predict whether the patient will benefit from operative or non-operative treatment. The classification system appears well considered; however, the classification needs validation and to be correlated to outcome.

Barfod et al. have developed a method for measuring the prolongation of the Achilles tendon in the acute phase following a rupture. The length measurement has been validated using healthy subjects. Data are analyzed and publication is expected autumn 2013. It has not been tested whether the measurement works on torn Achilles tendons and whether there is a correlation between the measurement and outcome.

With this project the investigators wish to:

1. Teste the reproducibility of Amlang's ultrasound classification by examining the intra- and inter-rater reliability.
2. Investigate whether Amlang's ultrasound classification is able to predict which patients are likely to develop complications when treated non-operatively.
3. Investigate whether Barfod's length measurement is able to predict which patients are likely to develop complications when treated non-operatively.

Study Design Type of study The study is carried out as a prospective cohort study. Time schedule The recruitment of patients will begin 1 of November 2013. It is expected that the study will be completed after 4-5 years; the recruitment itself is expected to span 2 years, provided that an average of 6 patients is included per month.

Discontinuation Each patient can choose to withdraw from the trial at any time. A patient may also be withdrawn from the trial at any time based on the investigators' discretion.

Method Amlang's ultrasound classification and Barfod's length measurement are determined as described below. For the initial 30 patients Amlang's ultrasound classification will be determined using two independent ultrasound-operators in order to test the inter-observer consistency.

Ultrasound - Set up The patient is in the prone position with the knees slightly flexed (10 -20 degrees). A triangular foam pad is placed below (anterior to) the ankle joints, so that the feet are resting limply. By moving the pad up (cranial) and down (caudal) the angle of the relaxed ankle joints is adjusted to 20 degrees plantar flexion. The angle is measured using a goniometer (the longitudinal axis of the fibula is at 110 degrees with the posterior part of the lateral border of the foot). The calf muscles are relaxed.

Amlang's ultrasound classification Amlang's ultrasound classification is conducted by determining the cross-sectional area of the widest point of the tendon below (distal to) the rupture (area-widest) and of the narrowest point at the rupture site (area-smallest). The ratio between "area-smallest" and "area-widest" is interpreted as a measure for the magnitude of overlap between the tendon ends. A ratio above 70 percent is considered as a total adaption of the tendon ends. A ratio of 30 to 70 percent is considered as a partial adaption of the tendon ends. And a ratio of less than 30 percent is considered as a lack of adaption of the tendon ends.

Barfod's length measurement Barfod's length measurement is conducted using a simple method that does not require expensive equipment or advanced instruments. A needle is placed between the skin and the ultrasonographic probe. The shadow of the needle then projects the internal structures to the skin surface and the distance between calcaneus and the medial head of the gastrocnemius muscle can then be measured.

Study Design Type of study The study is carried out as a prospective cohort study. Time schedule The recruitment of patients will begin 1 of November 2013. It is expected that the study will be completed after 4-5 years; the recruitment itself is expected to span 2 years, provided that an average of 6 patients is included per month.

Discontinuation Each patient can choose to withdraw from the trial at any time. A patient may also be withdrawn from the trial at any time based on the investigators' discretion.

Method Amlang's ultrasound classification and Barfod's length measurement are determined as described below. For the initial 30 patients Amlang's ultrasound classification will be determined using two independent ultrasound-operators in order to test the inter-observer consistency.

Ultrasound - Set up The patient is in the prone position with the knees slightly flexed (10 -20 degrees). A triangular foam pad is placed below (anterior to) the ankle joints, so that the feet are resting limply. By moving the pad up (cranial) and down (caudal) the angle of the relaxed ankle joints is adjusted to 20 degrees plantar flexion. The angle is measured using a goniometer (the longitudinal axis of the fibula is at 110 degrees with the posterior part of the lateral border of the foot). The calf muscles are relaxed.

Amlang's ultrasound classification Amlang's ultrasound classification is conducted by determining the cross-sectional area of the widest point of the tendon below (distal to) the rupture (area-widest) and of the narrowest point at the rupture site (area-smallest). The ratio between "area-smallest" and "area-widest" is interpreted as a measure for the magnitude of overlap between the tendon ends. A ratio above 70 percent is considered as a total adaption of the tendon ends. A ratio of 30 to 70 percent is considered as a partial adaption of the tendon ends. And a ratio of less than 30 percent is considered as a lack of adaption of the tendon ends.

Barfod's length measurement Barfod's length measurement is conducted using a simple method that does not require expensive equipment or advanced instruments. A needle is placed between the skin and the ultrasonographic probe. The shadow of the needle then projects the internal structures to the skin surface and the distance between calcaneus and the medial head of the gastrocnemius muscle can then be measured.

Statistics The groups will be described descriptively regarding demographic parameters as well as primary and secondary endpoints. The correlation between Amlang's ultrasound classification and the primary and secondary endpoints will be examined using a regression analysis. The correlation between Barfod's length measurement and the primary and secondary endpoints will be examined in the same way.

The research group The study is carried out as collaboration between the research unit, Clinical Orthopaedic Research Hvidovre (www.corh.dk) and the Department of Physical- and Occupational Therapy, both at Copenhagen University Hospital Hvidovre.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* The patient must be expected to be able to attend rehabilitation and post-examinations.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.

Exclusion Criteria:

* Former rupture of one or both Achilles tendon(s).
* Previous surgery on the Achilles tendon.
* Fluoroquinolone treatment within the last 6 months.
* Tendinosis treated with corticosteroids (tablets or injections) within the last 6 months.
* The patient has been diagnosed with arterial insufficiency in the legs.
* Terminal illness or severe medical illness: ASA score higher than or equal to 3.
* The space between the rupture and the calcaneus is less than 1cm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 patients who are treated for acute Achilles tendon rupture at Copenhagen University Hospital Hvidovre. Patients who fulfil the inclusion criteria but do not wish to participate are treated according the standard regimen (non-operatively without early controlled movement of the ankle joint).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Corelation between Amlangs ultrasound classification or Barfods length meassure and ATRS | 1 year
  We whish to investigate if Amlangs ultrasound classification or Barfods length meassure can predict outcome after acute achilles tendon rupture. To do so both meassures will be correlated to ATRS (the Achilles tendon Total Rupture Score).

SECONDARY OUTCOMES:
Correlation between Amlangs Ultrasound Classification or Barfods length meassure and Heel-rise-work test | 1 year
  We whish to investigate if Amlangs ultrasound classification or Barfods length meassure can predict outcome after acute achilles tendon rupture. To do so both meassures will be correlated to the heel-rise work test.
  Heel-rise-work test: Endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel-rises are counted and measured. The results are then compared to the weight of the patient and the total work is estimated. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used.

OTHER OUTCOMES:
Correlation between Amlangs Ultrasound Classification or Barfods length meassure and Re-rupture | 1 year
  We whish to investigate if Amlangs ultrasound classification or Barfods length meassure can predict outcome after acute achilles tendon rupture. To do so both meassures will be correlated to the rate of re-rupture.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark